CLINICAL TRIAL: NCT06373588
Title: Co-design and Evaluation of a Patient Navigator Intervention for Migrant Children and Youth with Special Healthcare Needs (CYSHCN) Experiencing Care Transitions (MiNav Trial)
Brief Title: Empowering Families of Migrant Children and Youth with Special Healthcare Needs
Acronym: MiNav
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Unity Health Toronto (Other); Canadian Institutes of Health Research (CIHR) (Other Government); The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Patricia Li, Associate Professor, Department of Pediatrics, Faculty of Medicine and Health Sciences, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MP-37-2023-9418
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-07

CONDITIONS: Patient Navigation
Keywords: Child Health; Chronic health diseases; Patient Navigation; Migrant population; Refugee; Immigrant; Asylum seeker; Culturally competent care; Health services research
MeSH Terms: interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: Multi-centre, pragmatic, assessor-blinded, parallel randomized controlled trial with an embedded qualitative study. In the control arm, participants will receive a standard information package and care usually provided within their clinics. In the intervention arm, participants will receive support from a trained patient navigator. The patient navigator will contact participants: 1) Within 7 days of randomization; 2) At least once every 3 months up to 12 months; 3) As needed to follow-up on tasks identified in previous visits; and 4) As initiated by the participant. The navigator will tailor the topics addressed during these interactions according to the needs of the participant and compile a care plan with input from the patient, family, and clinicians.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Participants will receive care usually provided within their clinics and a standard package with healthcare resources. In keeping with the pragmatic design, there will be variation in the support provided for navigation and care coordination, referral patterns to health and social services, as well as community resources. However, we will document these differences to provide context about potential differences in effects which may occur between sites.
- Patient Navigator (Experimental): Participants will be paired with a patient navigator. The patient navigator will contact participants: 1) Within 7 days of randomization; 2) At least once every 3 months up to 12 months; 3) As needed to follow-up on tasks identified in previous visits; and 4) As initiated by the participant. Contacts will occur during in-person clinic visits (prioritized for first encounter, if possible), or over video, telephone, SMS, and/or emails. The navigator will tailor the topics addressed during these interactions according to the needs of the participant and compile a care plan with input from the patient, family, and clinicians. In addition, to assess intervention fidelity, patient navigators will document all participant contacts on standardized forms, including topics addressed, services and coordination provided, written care plan provided, and concurrent resources/interventions accessed (e.g., social worker, funding/housing applications, support from community organizations).
  Interventions: Behavioral: Patient Navigator

INTERVENTIONS:
Behavioral: Patient Navigator — The patient navigator will meet the following requirements: a bachelor's degree in health or social sciences, or equivalent experiences; strong knowledge of the local health and social services system; trauma-informed care and cultural safety; strong interpersonal skills, ability to problem-solve, and autonomy; have prior experiences with migrant communities (including lived experiences) and working in healthcare setting. The navigator will be trained on topics related to their role, through case discussions, and role playing, as done in other navigator trials. Topics will include Indigenous cultural safety as applied to migrant health, systems navigation, care coordination, family-centred care, social determinants of health (health insurance, income supplements, etc.) and inequities, advanced communication and helping skills (e.g., motivational interviewing), ethics, privacy, and confidentiality, and others as determined through our co-design process.
  Arms: Patient Navigator

SUMMARY:
The goal of this randomized controlled trial is to test if a patient navigator program improves healthcare experiences and outcomes for migrant families caring for a child or youth with special healthcare needs (i.e. chronic health condition).

The main questions are, for migrant families with a child or youth with special healthcare needs:

Does a patient navigator reduces barriers to care? Does a patient navigator improve care coordination, caregiver empowerment, caregiver stress and quality of life? What are the healthcare experiences for families with and without the patient navigator intervention?

Participants will:

* Receive the intervention, i.e., the patient navigator program, or continue with standard of care for 12 months
* Fill out questionnaires at 3 time points on barriers to care, caregiver stress, care coordination, and their child's health

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of child/youth ≤18 years who is first- or second-generation migrant, defined as born outside of Canada or having parents born elsewhere, respectively (migrants include immigrants, resettled refugees, refugee claimants (asylum seekers), temporary workers or international students, and other individuals without formal immigration status (undocumented)).
* Children or youth with special health care needs, as defined by the CYSHCN Screener, which identifies children who are experiencing one or more functional limitation or service use due to a physical, emotional, behavioural, developmental, or other health condition that has lasted or is expected to last at least 12 months.
* Experiencing care transitions between at least 2 of the following: primary care, community-based care, secondary specialist care, and/or hospital-based (acute) care.

Exclusion Criteria:

* Caregiver living in Canada ≥10 years
* Families who are receiving available peer navigation support at sites will be excluded to limit cross-over of interventions.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 324 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Barriers to Care (BCQ) | Assessment will happen at baseline, 6 months after the start of the intervention and at the end of the intervention, i.e., 12 months.
  The BCQ has been validated for children and youth with special healthcare needs. It contains 39 items grouped in 5 sub-scales, which include: 1) Pragmatics: issues related to logistics and costs that may prevent or delay appropriate utilization; 2) Skills: strategies to navigate or function competently in health system care; 3) Expectations: caregiver expectations of receiving poor quality care, including a lack of communication between doctors, health care system; 4) Marginalization: the "internationalization and personalization of negative experiences within the health care system"; 5) Knowledge and beliefs: personal ideas about nature and treatment of illness (including culture), which may differ from the healthcare provider. Caregivers rate the items on a 5-point Likert scale, converted to a score ranging from 0 to 100 (higher scores = fewer barriers).

SECONDARY OUTCOMES:
Effective care coordination | Assessment will happen at baseline, 6 months after the start of the intervention and at the end of the intervention, i.e., 12 months.
  Based on 6 questions from the National Survey on children with special health care needs, as care coordination that is adequate (receiving help and satisfied), inadequate (not receiving and less than very satisfied), or no need for care coordination.
  The primary goals of this survey is to assess the impact of special health care needs and to evaluate change over time.
Parental empowerment scale | Assessment will happen at baseline, 6 months after the start of the intervention and at the end of the intervention, i.e., 12 months.
  A validated scale in families with children or youth with special healthcare needs. We will use the 12-item "Service System" subscale, which measures empowerment using a 5-point Likert scale converted to a score ranging from 1- 70 (higher scores = increased services) as it pertains to the caregiver actively working to get the services required for their child.
Healthcare utilization | Assessment will happen at baseline, 6 months after the start of the intervention and at the end of the intervention, i.e., 12 months.
  ER visits, hospital admissions, and no-show visits, through chart review and patient reports.
PROMIS - Pediatric Global Health 7 | Assessment will happen at baseline, 6 months after the start of the intervention and at the end of the intervention, i.e., 12 months.
  Parent-reported assessment of their child's perceived health, quality of life and physical/mental health using a 5-point likert scale. Converted to a score ranging from 1 to 20 (higher scores = better perceived health).
Short-form survey 12 | Assessment will happen at baseline, 6 months after the start of the intervention and at the end of the intervention, i.e., 12 months.
  For caregivers; This is a self-reported outcome measure that measures quality of life. This one question is scored from 1 poor health - 4 excellent health.
Patient Health Questionnaire (PHQ-2) | Assessment will happen at baseline, 6 months after the start of the intervention and at the end of the intervention, i.e., 12 months.
  For caregivers; The PHQ-2 inquires about the frequency of depressed mood and anhedonia over the past two weeks. This questionnaire is used to screen for depression in a "first-step" approach. The PHQ-2 score ranges from 0-6 with a score higher than 3 indicating a likelihood of depression.
Distress Thermometer | Assessment will happen at baseline, 6 months after the start of the intervention and at the end of the intervention, i.e., 12 months.
  The distress thermometer asks participants their level of distress in the past month on a scale of 0-10, 10 indicating extreme distress.
Perceived stress scale | Assessment will happen at baseline, 6 months after the start of the intervention and at the end of the intervention, i.e., 12 months.
  10-item scale designed to help measure individual stress levels in various situations. PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Patient Satisfaction with Interpersonal Relationships with Navigators (PSN-I) | Assessment will happen at 6 months and at the end of the intervention, i.e., 12 months, only for the intervention group.
  A valid and reliable measure of satisfaction with patient navigators that contains 9-item answered with a 5-point Likert scale. Score ranging from 1- 45, higher score reflects higher satisfaction with patient navigator.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Li, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (3):
- Canada (3):
  - Unity Health Toronto, Compass Clinic, Toronto, Ontario
  - CIUSSS West-Central Montreal, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McPherson M, Arango P, Fox H, Lauver C, McManus M, Newacheck PW, Perrin JM, Shonkoff JP, Strickland B. A new definition of children with special health care needs. Pediatrics. 1998 Jul;102(1 Pt 1):137-40. doi: 10.1542/peds.102.1.137. No abstract available. PMID 9714637
- [Background] Arim RG, Kohen DE, Brehaut JC, Guevremont A, Garner RE, Miller AR, McGrail K, Brownell M, Lach LM, Rosenbaum PL. Developing a non-categorical measure of child health using administrative data. Health Rep. 2015 Feb;26(2):9-16. PMID 25692939
- [Background] Antonelli R, McAllister J, Popp J. Making Care Coordination a Critical Component of the Pediatric Health System: A Multidisciplinary Framework. 2009.
- [Background] Cordeiro A, Davis RK, Antonelli R, Rosenberg H, Kim J, Berhane Z, Turchi R. Care Coordination for Children and Youth With Special Health Care Needs: National Survey Results. Clin Pediatr (Phila). 2018 Oct;57(12):1398-1408. doi: 10.1177/0009922818783501. Epub 2018 Jun 22. PMID 29932000
- [Background] Fox F, Aabe N, Turner K, Redwood S, Rai D. "It was like walking without knowing where I was going": A Qualitative Study of Autism in a UK Somali Migrant Community. J Autism Dev Disord. 2017 Feb;47(2):305-315. doi: 10.1007/s10803-016-2952-9. PMID 27858263
- [Background] Khanlou N, Haque N, Sheehan S, Jones G. "It is an Issue of not Knowing Where to Go": Service Providers' Perspectives on Challenges in Accessing Social Support and Services by Immigrant Mothers of Children with Disabilities. J Immigr Minor Health. 2015 Dec;17(6):1840-7. doi: 10.1007/s10903-014-0122-8. PMID 25376126
- [Background] Alsharaydeh EA, Alqudah M, Lee RLT, Chan SW. Challenges, Coping, and Resilience Among Immigrant Parents Caring for a Child With a Disability: An Integrative Review. J Nurs Scholarsh. 2019 Nov;51(6):670-679. doi: 10.1111/jnu.12522. Epub 2019 Oct 21. PMID 31637861
- [Background] Yu SM, Singh GK. Household language use and health care access, unmet need, and family impact among CSHCN. Pediatrics. 2009 Dec;124 Suppl 4:S414-9. doi: 10.1542/peds.2009-1255M. PMID 19948607
- [Background] Son E, Moring NS, Igdalsky L, Parish SL. Navigating the health-care system in community: Perspectives from Asian immigrant parents of children with special health-care needs. J Child Health Care. 2018 Jun;22(2):251-268. doi: 10.1177/1367493517753084. Epub 2018 Jan 28. PMID 29374977
- [Background] Kalich A, Heinemann L, Ghahari S. A Scoping Review of Immigrant Experience of Health Care Access Barriers in Canada. J Immigr Minor Health. 2016 Jun;18(3):697-709. doi: 10.1007/s10903-015-0237-6. PMID 26093784
- [Background] Salami B, Mason A, Salma J, Yohani S, Amin M, Okeke-Ihejirika P, Ladha T. Access to Healthcare for Immigrant Children in Canada. Int J Environ Res Public Health. 2020 May 10;17(9):3320. doi: 10.3390/ijerph17093320. PMID 32397618
- [Background] Ahmed S, Shommu NS, Rumana N, Barron GR, Wicklum S, Turin TC. Barriers to Access of Primary Healthcare by Immigrant Populations in Canada: A Literature Review. J Immigr Minor Health. 2016 Dec;18(6):1522-1540. doi: 10.1007/s10903-015-0276-z. PMID 26364053
- [Background] McKeary M, Newbold B. Barriers to care: the challenges for Canadian refugees and their health care providers. Journal of Refugee Studies. 2010;23(4):523-545.
- [Background] Campbell RM, Klei AG, Hodges BD, Fisman D, Kitto S. A comparison of health access between permanent residents, undocumented immigrants and refugee claimants in Toronto, Canada. J Immigr Minor Health. 2014 Feb;16(1):165-76. doi: 10.1007/s10903-012-9740-1. PMID 23124632
- [Background] Woodgate RL, Busolo DS, Crockett M, Dean RA, Amaladas MR, Plourde PJ. A qualitative study on African immigrant and refugee families' experiences of accessing primary health care services in Manitoba, Canada: it's not easy! Int J Equity Health. 2017 Jan 9;16(1):5. doi: 10.1186/s12939-016-0510-x. PMID 28068998
- [Background] McLeroy KR, Bibeau D, Steckler A, Glanz K. An ecological perspective on health promotion programs. Health Educ Q. 1988 Winter;15(4):351-77. doi: 10.1177/109019818801500401. PMID 3068205
- [Background] Tirado V, Chu J, Hanson C, Ekstrom AM, Kagesten A. Barriers and facilitators for the sexual and reproductive health and rights of young people in refugee contexts globally: A scoping review. PLoS One. 2020 Jul 20;15(7):e0236316. doi: 10.1371/journal.pone.0236316. eCollection 2020. PMID 32687519
- [Background] Arfa S, Solvang PK, Berg B, Jahnsen R. Disabled and immigrant, a double minority challenge: a qualitative study about the experiences of immigrant parents of children with disabilities navigating health and rehabilitation services in Norway. BMC Health Serv Res. 2020 Feb 22;20(1):134. doi: 10.1186/s12913-020-5004-2. PMID 32087730
- [Background] Yaseen W, Steckle V, Sgro M, Barozzino T, Suleman S. Exploring Stakeholder Service Navigation Needs for Children with Developmental and Mental Health Diagnoses. J Dev Behav Pediatr. 2021 Sep 1;42(7):553-560. doi: 10.1097/DBP.0000000000000924. PMID 34518497
- [Background] Dimitropoulos G, Morgan-Maver E, Allemang B, Schraeder K, Scott SD, Pinzon J, Andrew G, Guilcher G, Hamiwka L, Lang E, McBrien K, Nettel-Aguirre A, Pacaud D, Zwaigenbaum L, Mackie A, Samuel S. Health care stakeholder perspectives regarding the role of a patient navigator during transition to adult care. BMC Health Serv Res. 2019 Jun 17;19(1):390. doi: 10.1186/s12913-019-4227-6. PMID 31208417
- [Background] Dundaru-Bandi D, Daianska A, Ferkli M, Morantz G, Li P. Addressing and Evaluating the Healthcare Needs of Refugee and Immigrant Families During the COVID-19 Pandemic. presented at: Pediatric Academic Society Meeting; 2021; Virtual (due to COVID).
- [Background] McBrien KA, Ivers N, Barnieh L, Bailey JJ, Lorenzetti DL, Nicholas D, Tonelli M, Hemmelgarn B, Lewanczuk R, Edwards A, Braun T, Manns B. Patient navigators for people with chronic disease: A systematic review. PLoS One. 2018 Feb 20;13(2):e0191980. doi: 10.1371/journal.pone.0191980. eCollection 2018. PMID 29462179
- [Background] Pedersen A, Hack TF. Pilots of oncology health care: a concept analysis of the patient navigator role. Oncol Nurs Forum. 2010 Jan;37(1):55-60. doi: 10.1188/10.ONF.55-60. PMID 20044339
- [Background] Wells KJ, Battaglia TA, Dudley DJ, Garcia R, Greene A, Calhoun E, Mandelblatt JS, Paskett ED, Raich PC; Patient Navigation Research Program. Patient navigation: state of the art or is it science? Cancer. 2008 Oct 15;113(8):1999-2010. doi: 10.1002/cncr.23815. PMID 18780320
- [Background] Shommu NS, Ahmed S, Rumana N, Barron GR, McBrien KA, Turin TC. What is the scope of improving immigrant and ethnic minority healthcare using community navigators: A systematic scoping review. Int J Equity Health. 2016 Jan 15;15:6. doi: 10.1186/s12939-016-0298-8. PMID 26768130
- [Background] Newacheck PW, Strickland B, Shonkoff JP, Perrin JM, McPherson M, McManus M, Lauver C, Fox H, Arango P. An epidemiologic profile of children with special health care needs. Pediatrics. 1998 Jul;102(1 Pt 1):117-23. doi: 10.1542/peds.102.1.117. PMID 9651423
- [Background] Lindsay S, King G, Klassen AF, Esses V, Stachel M. Working with immigrant families raising a child with a disability: challenges and recommendations for healthcare and community service providers. Disabil Rehabil. 2012;34(23):2007-17. doi: 10.3109/09638288.2012.667192. Epub 2012 Mar 29. PMID 22455458
- [Background] Banerjee AT, Watt L, Gulati S, Sung L, Dix D, Klassen R, Klassen AF. Cultural beliefs and coping strategies related to childhood cancer: the perceptions of South Asian immigrant parents in Canada. J Pediatr Oncol Nurs. 2011 May-Jun;28(3):169-78. doi: 10.1177/1043454211408106. Epub 2011 Jun 6. PMID 21646638
- [Background] Tuyisenge G, Goldenberg SM. COVID-19, structural racism, and migrant health in Canada. Lancet. 2021 Feb 20;397(10275):650-652. doi: 10.1016/S0140-6736(21)00215-4. Epub 2021 Feb 1. No abstract available. PMID 33539727
- [Background] Bradby H, Varyani M, Oglethorpe R, Raine W, White I, Helen M. British Asian families and the use of child and adolescent mental health services: a qualitative study of a hard to reach group. Soc Sci Med. 2007 Dec;65(12):2413-24. doi: 10.1016/j.socscimed.2007.07.025. Epub 2007 Sep 4. PMID 17766019
- [Background] Narayan N. Interplay between cultural beliefs and attitudes in raising a child with Intellectual Disability-An Asian Indian Study. Alliant International University; 2014.
- [Background] Jegatheesan B. Muslim children with autism learn to pray. J Dev Behav Pediatr. 2010 Jun;31(5):458-9. doi: 10.1097/DBP.0b013e3181d59470. No abstract available. PMID 20535085
- [Background] King G, Desmarais C, Lindsay S, Pierart G, Tetreault S. The roles of effective communication and client engagement in delivering culturally sensitive care to immigrant parents of children with disabilities. Disabil Rehabil. 2015;37(15):1372-81. doi: 10.3109/09638288.2014.972580. Epub 2014 Oct 17. PMID 25323397
- [Background] Browne AJ, Varcoe C, Ward C. San'yas Indigenous Cultural Safety Training as an educational intervention: Promoting anti-racism and equity in health systems, policies, and practices. The International Indigenous Policy Journal. 2021;12(3):1-26.
- [Background] Osei-Twum J, Puffer E, Banerjee AT. Indigenous Cultural Safety: Exploring The Applicability Of The Concepts To Immigrant Health Care. In Bruce Newbold & Kathi Wilson (Eds.), A Research Agenda for Migration and Health. 1st ed. Edward Elgar; 2019.
- [Background] Curtis E, Jones R, Tipene-Leach D, Walker C, Loring B, Paine SJ, Reid P. Why cultural safety rather than cultural competency is required to achieve health equity: a literature review and recommended definition. Int J Equity Health. 2019 Nov 14;18(1):174. doi: 10.1186/s12939-019-1082-3. PMID 31727076
- [Background] Brown A, McIsaac J-L, Reddington S, et al. Newcomer families' experiences with programs and services to support early childhood development in Canada: A scoping review. Journal of Childhood, Education & Society. 2020;1(2)
- [Background] John A, Bower K, McCullough S. Indian immigrant parents of children with developmental disabilities: stressors and support systems. Early Child Development and Care. 2016;186(10)
- [Background] Peart A, Lewis V, Brown T, Russell G. Patient navigators facilitating access to primary care: a scoping review. BMJ Open. 2018 Mar 17;8(3):e019252. doi: 10.1136/bmjopen-2017-019252. PMID 29550777
- [Background] Luke A, Doucet S, Azar R. Paediatric patient navigation models of care in Canada: An environmental scan. Paediatr Child Health. 2018 May;23(3):e46-e55. doi: 10.1093/pch/pxx176. Epub 2018 Jan 2. PMID 29769815
- [Background] Frakking TT, Teoh HJ, Shelton D, Moloney S, Ward D, Annetts K, David M, Levitt D, Chang AB, Carty C, Barber M, Carter HE, Mickan S, Weir KA, Waugh J. Effect of Care Coordination Using an Allied Health Liaison Officer for Chronic Noncomplex Medical Conditions in Children: A Multicenter Randomized Clinical Trial. JAMA Pediatr. 2022 Mar 1;176(3):244-252. doi: 10.1001/jamapediatrics.2021.5465. PMID 34962514
- [Background] Merariu J, Sabsabi B, Ferkli M, Li P. Evaluating a Newcomer Navigator Program for the Montreal Children's Hospital Multicultural Clinic. presented at: North American Refugee Health Conference; 2021; Virtual (due to COVID).
- [Background] Suleman S, Milone F, Rollins M, Vojvoda D, Barozzino T. Implementation of a pediatric patient navigator for children with developmetnal or mental health concerns. Paediatrics & Child Health. 2018;23(1):e56.
- [Background] Arya N, Redditt VJ, Talavlikar R, Holland T, Brindamour M, Wright V, Saad A, Beukeboom C, Coakley A, Rashid M, Pottie K. Caring for refugees and newcomers in the post-COVID-19 era: Evidence review and guidance for FPs and health providers. Can Fam Physician. 2021 Aug;67(8):575-581. doi: 10.46747/cfp.6708575. PMID 34385202
- [Background] Rizwan A, Suleman S. An Evidence-Based Model of Care for Newcomer Children with Special Health Care Needs. Paediatrics & Child Health. 2020;25(2):e47-48.
- [Background] Greenhalgh T, Jackson C, Shaw S, Janamian T. Achieving Research Impact Through Co-creation in Community-Based Health Services: Literature Review and Case Study. Milbank Q. 2016 Jun;94(2):392-429. doi: 10.1111/1468-0009.12197. PMID 27265562
- [Background] Moll S, Wyndham-West M, Mulvale G, Park S, Buettgen A, Phoenix M, Fleisig R, Bruce E. Are you really doing 'codesign'? Critical reflections when working with vulnerable populations. BMJ Open. 2020 Nov 3;10(11):e038339. doi: 10.1136/bmjopen-2020-038339. PMID 33148733
- [Background] Turchi RM, Berhane Z, Bethell C, Pomponio A, Antonelli R, Minkovitz CS. Care coordination for CSHCN: associations with family-provider relations and family/child outcomes. Pediatrics. 2009 Dec;124 Suppl 4:S428-34. doi: 10.1542/peds.2009-1255O. PMID 19948609
- [Background] Bethell CD, Read D, Stein RE, Blumberg SJ, Wells N, Newacheck PW. Identifying children with special health care needs: development and evaluation of a short screening instrument. Ambul Pediatr. 2002 Jan-Feb;2(1):38-48. doi: 10.1367/1539-4409(2002)0022.0.co;2. PMID 11888437
- [Background] Seid M, Sobo EJ, Gelhard LR, Varni JW. Parents' reports of barriers to care for children with special health care needs: development and validation of the barriers to care questionnaire. Ambul Pediatr. 2004 Jul-Aug;4(4):323-31. doi: 10.1367/A03-198R.1. PMID 15264959
- [Background] Borm GF, Fransen J, Lemmens WA. A simple sample size formula for analysis of covariance in randomized clinical trials. J Clin Epidemiol. 2007 Dec;60(12):1234-8. doi: 10.1016/j.jclinepi.2007.02.006. Epub 2007 Jun 6. PMID 17998077
- [Background] Samuel S, Dimitropoulos G, Schraeder K, Klarenbach S, Nettel-Aguirre A, Guilcher G, Pacaud D, Pinzon J, Lang E, Andrew G, Zwaigenbaum L, Scott S, McBrien K, Hamiwka L, Mackie A. Pragmatic trial evaluating the effectiveness of a patient navigator to decrease emergency room utilisation in transition age youth with chronic conditions: the Transition Navigator Trial protocol. BMJ Open. 2019 Dec 10;9(12):e034309. doi: 10.1136/bmjopen-2019-034309. PMID 31826899
- [Background] Bender JL, Flora PK, Milosevic E, Soheilipour S, Maharaj N, Dirlea M, Parvin L, Matthew A, Kazanjian A. Training prostate cancer survivors and caregivers to be peer navigators: a blended online/in-person competency-based training program. Support Care Cancer. 2021 Mar;29(3):1235-1244. doi: 10.1007/s00520-020-05586-8. Epub 2020 Jul 2. PMID 32613373
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318
- [Background] Seid M, Opipari-Arrigan L, Gelhard LR, Varni JW, Driscoll K. Barriers to care questionnaire: reliability, validity, and responsiveness to change among parents of children with asthma. Acad Pediatr. 2009 Mar-Apr;9(2):106-13. doi: 10.1016/j.acap.2008.12.003. Epub 2009 Feb 11. PMID 19329101
- [Background] Koren PE, DeChillo N, Friesen BJ. Measuring empowerment in families whose children have emotional disabilities: A brief questionnaire. Rehabilitation Psychology. 1992;37(4):305-321.
- [Background] Segers EW, van den Hoogen A, van Eerden IC, Hafsteinsdottir T, Ketelaar M. Perspectives of parents and nurses on the content validity of the Family Empowerment Scale for parents of children with a chronic condition: A mixed-methods study. Child Care Health Dev. 2019 Jan;45(1):111-120. doi: 10.1111/cch.12629. PMID 30426545
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Baik SH, Fox RS, Mills SD, Roesch SC, Sadler GR, Klonoff EA, Malcarne VL. Reliability and validity of the Perceived Stress Scale-10 in Hispanic Americans with English or Spanish language preference. J Health Psychol. 2019 Apr;24(5):628-639. doi: 10.1177/1359105316684938. Epub 2017 Jan 5. PMID 28810432
- [Background] Bastianon CD, Klein EM, Tibubos AN, Brahler E, Beutel ME, Petrowski K. Perceived Stress Scale (PSS-10) psychometric properties in migrants and native Germans. BMC Psychiatry. 2020 Sep 11;20(1):450. doi: 10.1186/s12888-020-02851-2. PMID 32917170
- [Background] Huang F, Wang H, Wang Z, Zhang J, Du W, Su C, Jia X, Ouyang Y, Wang Y, Li L, Jiang H, Zhang B. Psychometric properties of the perceived stress scale in a community sample of Chinese. BMC Psychiatry. 2020 Mar 20;20(1):130. doi: 10.1186/s12888-020-02520-4. PMID 32197589
- [Background] Kim HJ. Reliability and Validity of the 4-Item Version of the Korean Perceived Stress Scale. Res Nurs Health. 2016 Dec;39(6):472-479. doi: 10.1002/nur.21745. Epub 2016 Aug 22. PMID 27546692
- [Background] Martynowska K, Korulczyk T, Mamcarz PJ. Perceived stress and well-being of Polish migrants in the UK after Brexit vote. PLoS One. 2020 Jul 23;15(7):e0236168. doi: 10.1371/journal.pone.0236168. eCollection 2020. PMID 32702031
- [Background] Nordin M, Nordin S. Psychometric evaluation and normative data of the Swedish version of the 10-item perceived stress scale. Scand J Psychol. 2013 Dec;54(6):502-7. doi: 10.1111/sjop.12071. Epub 2013 Oct 5. PMID 24118069
- [Background] Remor E. Psychometric properties of a European Spanish version of the Perceived Stress Scale (PSS). Span J Psychol. 2006 May;9(1):86-93. doi: 10.1017/s1138741600006004. PMID 16673626
- [Background] Ravens-Sieberer U, Gosch A, Rajmil L, Erhart M, Bruil J, Power M, Duer W, Auquier P, Cloetta B, Czemy L, Mazur J, Czimbalmos A, Tountas Y, Hagquist C, Kilroe J; KIDSCREEN Group. The KIDSCREEN-52 quality of life measure for children and adolescents: psychometric results from a cross-cultural survey in 13 European countries. Value Health. 2008 Jul-Aug;11(4):645-58. doi: 10.1111/j.1524-4733.2007.00291.x. Epub 2007 Dec 17. PMID 18179669
- [Background] Jean-Pierre P, Shao C, Cheng Y, Wells KJ, Paskett E, Fiscella K. Patient Satisfaction with Navigator Interpersonal Relationship (PSN-I): item-level psychometrics using IRT analysis. Support Care Cancer. 2020 Feb;28(2):541-550. doi: 10.1007/s00520-019-04833-x. Epub 2019 May 10. PMID 31076896
- [Background] Charmaz K. Constructing grounded theory. 2nd edition ed. Introducing qualitative methods. Sage; 2014:xxi, 388 pages.
- [Background] Klassen AF, Gulati S, Watt L, Banerjee AT, Sung L, Klaassen RJ, Dix D, Poureslami IM, Shaw N. Immigrant to Canada, newcomer to childhood cancer: a qualitative study of challenges faced by immigrant parents. Psychooncology. 2012 May;21(5):558-62. doi: 10.1002/pon.1963. Epub 2011 Mar 21. PMID 21425390
- [Background] Davis K, Minckas N, Bond V, Clark CJ, Colbourn T, Drabble SJ, Hesketh T, Hill Z, Morrison J, Mweemba O, Osrin D, Prost A, Seeley J, Shahmanesh M, Spindler EJ, Stern E, Turner KM, Mannell J. Beyond interviews and focus groups: a framework for integrating innovative qualitative methods into randomised controlled trials of complex public health interventions. Trials. 2019 Jun 6;20(1):329. doi: 10.1186/s13063-019-3439-8. PMID 31171041
- [Background] Cresswell JW, Poth CN. Qualitative Inquiry & Research Design: Choosing among five approaches. 6th ed. 2018.
- [Background] Charmaz K. The Power of Constructivist Grounded Theory for Critical Inquiry. Qualitative Inquiry. 2017;23(1):34-45. doi:10.1177/1077800416657105
- [Background] Guruge S, Khanlou N. Intersectionalities of influence: researching the health of immigrant and refugee women. Can J Nurs Res. 2004 Sep;36(3):32-47. PMID 15551661
- [Background] Spradley JP. The ethnographic interview. Holt, Rinehart and Winston; 1979:vii, 247 p.
- [Background] Williamson DL, Choi J, Charchuk M, et al. Interpreter-facilitated cross-language interviews: a research note. Qualitative research. 2011;11(4):381-94.
- [Background] Elo S, Kyngas H. The qualitative content analysis process. J Adv Nurs. 2008 Apr;62(1):107-15. doi: 10.1111/j.1365-2648.2007.04569.x. PMID 18352969
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Impact of the South Asian Adolescent Diabetes Awareness Program (SAADAP) on diabetes knowledge, risk perception and health behaviour.
- [Background] Weidman DR, Desmarais P, Stevens K, Klinger CA, Colquhoun H, Bender JL, Gupta A. Peer Support Needs of Adolescents with Cancer in Pediatrics: A Canadian Mixed Methods Study. J Adolesc Young Adult Oncol. 2022 Aug;11(4):433-438. doi: 10.1089/jayao.2021.0122. Epub 2021 Sep 30. PMID 34591689
- [Background] McKay S. Immigrant Children With Special Health Care Needs: A Review. Curr Probl Pediatr Adolesc Health Care. 2019 Feb;49(2):45-49. doi: 10.1016/j.cppeds.2019.01.004. Epub 2019 Feb 15. PMID 30777710
- [Background] Merry L, Pelaez S. Knowledge translation and better health and health care for migrants in Canada: What is the responsibility of health funders and researchers? Can Fam Physician. 2021 Jun;67(6):403-405. doi: 10.46747/cfp.6706403. No abstract available. PMID 34127460
- See also: United States Census Bureau. 2020 National Survey of Children's Health. Accessed December 31, 2021 — https://www2.census.gov/programs-surveys/nsch/technical-documentation/codebook/NSCH_2020_Screener_Frequencies.pdf
- See also: Canadian Institutes of Health Research. (2021). Transitions in Care. Retrieved from Government of Canada: Canadian Institutes of Health Research. Accessed December 30, 2022 — https://cihr-irsc.gc.ca/e/50972.html
- See also: Children with an immigrant background: Bridging cultures — http://www12.statcan.gc.ca/census-recensement/2016/as-sa/98-200-x/2016015/98-200-x2016015-eng.cfm
- See also: Statistics Canada. Social Assistance Receipt Among Refugee Claimants in Canada — http://www150.statcan.gc.ca/n1/pub/11-626-x/11-626-x2015051-eng.htm
- See also: Social Planning Toronto. Unequal City: The Hidden Divide Among Toronto's Children and Youth — http://www.socialplanningtoronto.org/unequal_city_the_hidden_divide_among_toronto_s_children_and_youth
- See also: National Care Coordination Standards for Children and Youth with Special Health Care Needs. — http://www.nashp.org/wp-content/uploads/2020/10/care-coordination-report-v5.pdf
- See also: Guidance on co-producing a research project. — http://www.invo.org.uk/wp-content/uploads/2019/04/Copro_Guidance_Feb19.pdf
- See also: WHO guidelines on hand hygiene in health care. — http://www.ncbi.nlm.nih.gov/books/NBK144013/pdf/Bookshelf_NBK144013.pdf
- See also: Geographic distribution of immigrants and recent immigrants and their proportion within the population of census metropolitan areas, Canada — http://www150.statcan.gc.ca/n1/daily-quotidien/171025/t001b-eng.htm#fn02
- See also: National Newcomer Navigation Network — http://www.newcomernavigation.ca/en/index.aspx